CLINICAL TRIAL: NCT01292200
Title: A RCT to Promote Mammography Adherence Among Chinese Immigrant Women
Brief Title: Breast Health in Chinese American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Temple University (Other); University of California, Los Angeles (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Judy Wang, Associate Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2010-185; R01CA142941-01A1 (NIH)
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Chinese women; Mammography; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- watch DVD and small group discussion (Experimental): Participants will watch the video in a group and discuss the video.
  Interventions: Behavioral: watch DVD and small group discussion
- watch video only (Placebo Comparator): watch a 22 minutes long video at home by herself.
  Interventions: Behavioral: watch DVD

INTERVENTIONS:
Behavioral: watch DVD and small group discussion — Women in the small-group discussion mode will be called by their community educators to determine possible dates, times, and places for group meetings. The small group sessions will be conducted near the participants' homes. Each small-group will consist of 5-10 participants who will first view a 20-minute video together and then discuss the content of the video as well as their barriers to screening for about 30 minutes. A community educator and an RA at the study site will facilitate the discussion in Chinese languages according to a structured guide.
  Arms: watch DVD and small group discussion
Behavioral: watch DVD — Women in the single video mode will receive a cultural video along with an information sheet on local free and low-cost screening programs by mail.
  Arms: watch video only

SUMMARY:
This four-and-a-half-year study will test the efficacy of viewing a theoretically based and culturally sensitive video followed by group discussion (vs. single viewing) in increasing mammography use. The results of this study will lead cancer control efforts to effectively decrease breast cancer screening disparities experienced by Chinese-America women.

DETAILED DESCRIPTION:
We will conduct a 4.5-year community-based RCT to study the impact of intervention approaches (small-group video discussion vs. single video mode) on mammography used among Chinese immigrant women. The small-group video discussion will be led by trained Chinese community health educators and trained bilingual research staff using a standardized structured protocol at all sites. In the single video mode, we will mail the intervention materials to women to view and/or read at home. We will recruit 974 Chinese women through our strong and well-established Chinese community partnerships in the metropolitan areas of Washington, DC (Lead PI: Dr. Judy Wang, Georgetown University-GU), New York (Site PI: Dr. Grace Ma at Temple University), and southern California (Site PI: Dr. Annette Maxwell, University of California, Los Angeles-UCLA). Participants' eligibility are listed under "eligibility criteria". We will not enroll US-born Chinese women as they are least likely to face cultural and language barriers to mammography and less likely to engage in our small-group discussion, which will be conducted in Chinese languages. Also, we will not enroll short-term visitors as our study involves four interviews over a 2-year period.

ELIGIBILITY:
Inclusion Criteria:

1. First generation Chinese women
2. Aged 42 and older
3. Have not had a mammogram in the past 2 years
4. Have never had breast cancer
5. Lived in the metropolitan DC, southern CA, and NY suburb; AND
6. Have no mammography screening scheduled in the next 6 month from time of enrollment

Exclusion Criteria:

1. Short-term visitors
2. US-born Chinese Americans

Min Age: 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 954 (Actual)
Dates: Start 2010-07; Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
3rd interview about receipt of mammography screening | 6-month post-intervention
  Measure the effect of small group video discussion on mammography screening adherence.

SECONDARY OUTCOMES:
4th interview about receipt of mammography screening | 21-month post-intervention
  Measure the effect of small group video discussion on repeated mammography screening adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Judy (Huei-Yu) Wang, Ph.D., Principal Investigator — Georgetown University
Locations (3):
- United States (3):
  - UCLA, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang JH, Mandelblatt JS, Liang W, Yi B, Ma IJ, Schwartz MD. Knowledge, cultural, and attitudinal barriers to mammography screening among nonadherent immigrant Chinese women: ever versus never screened status. Cancer. 2009 Oct 15;115(20):4828-38. doi: 10.1002/cncr.24517. PMID 19645031
- [Background] Wang JH, Liang W, Schwartz MD, Lee MM, Kreling B, Mandelblatt JS. Development and evaluation of a culturally tailored educational video: changing breast cancer-related behaviors in Chinese women. Health Educ Behav. 2008 Dec;35(6):806-20. doi: 10.1177/1090198106296768. Epub 2007 Jun 29. PMID 17602099
- [Derived] Tan NQP, Ma GX, Maxwell AE, Brown RL, Zhou K, Loh A, Young L, Volk RJ, Lu Q, Wang JH. The impact of a small-group mammography video discussion on promoting screening uptake among nonadherent Chinese American immigrant women: A randomized controlled trial. Cancer. 2025 Jan 1;131(1):e35524. doi: 10.1002/cncr.35524. Epub 2024 Sep 10. PMID 39257218